CLINICAL TRIAL: NCT02240277
Title: Meropenem and Ciprofloxacin Dosing in the Critically Ill Patient With Septic Shock - a Single Center Pharmacokinetic Study
Brief Title: Meropenem and Ciprofloxacin Dosing in Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: The University of Queensland (Other)
Responsible Party: Principal Investigator, Fredrik Sjövall, MD, PhD, Rigshospitalet, Denmark
Other Study IDs: RH-RBWH-2014-1; 2014-002555-26 (EudraCT Number)
Record Dates: First submitted 2014-09-05; First posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Septic Shock
Keywords: Septic Shock; Meropenem; Ciprofloxacin; Pharmacokinetics
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with septic shock may have altered volume of distribution and metabolism of antibiotics which are crucial medications for treating infections. The aim of the study is to investigate the blood concentrations of Meropenem and Ciprofloxacin, two commonly used antibiotics, in patients with septic shock. The hypothesis is that standard dosing may produce insufficient levels of antibiotics in patients with septic shock.

DETAILED DESCRIPTION:
Sepsis may induce changes in renal function, increased capillary leakage and frequently blood-flow stasis in the peripheral tissues leading to an increase in the water space and diffusion distances. Significant changes have been observed in the distribution volume of certain antibiotics in patients with sepsis. The increased volume of distribution of water-soluble drugs is caused by a capillary leak syndrome that results in a net movement of fluid from the intravascular compartment into tissues. This capillary leak syndrome has been well described in patients with sepsis and may result in low trough serum concentrations. This, in turn, may result in a slow antibiotic penetration of tissues and a low tissue antibiotic concentration. Treatment failure may result if antibiotic choice or doses are incorrect and there is a lack of information which describes how to alter drug dosing in response to this increased volume of distribution in sepsis. Previous research has shown that some intensive care unit (ICU) patients have larger than normal between subject variability in drug clearance and volumes that can be attributed to supranormal renal clearances.

Aims of the present study:

1. To evaluate present meropenem and ciprofloxacin dosing and achieved plasma concentrations in relation to bacterial susceptibility.
2. To evaluate how to accurately dose meropenem and ciprofloxacin in patients with sepsis The overall hypothesis for this project is that some patients admitted to ICU with severe sepsis are undertreated with meropenem and ciprofloxacin using the dosing based on that recommended by the Product Information

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <90 years
* Clinical indication for therapy of one of the study antibiotics Meropenem or Ciprofloxacin in patients diagnosed at or during admission to ICU with septic shock
* Sepsis will be defined as:

  * Clinical suspicion of infection and/or Positive culture results
  * Systemic inflammatory response syndrome (SIRS) as defined by 2 or more of the following:
  * Core temperature < 36o C or > 38o C
  * Tachycardia as defined by a heart rate > 90 beats per minute
  * Tachypnoea as defined by a respiratory rate greater than 20 breaths per minute OR a PaCO2 less than 32 mmHg during spontaneous ventilation OR the requirement for mechanical ventilation.
  * A white blood cell count > 12 X 109 / L OR < 4 X 109 / L OR greater than 10 % immature (band) forms.
* Septic shock will be defined as:

  * Sepsis with persistent hypotension, systolic blood pressure < 90 mmHg or mean arterial pressure < 65 despite adequate fluid resuscitation
  * Requirement of inotropic support.
* Normal renal function as defined by:

  * Serum creatinine <170 mmol/L

Exclusion Criteria:

* Pre-existing renal impairment as defined by:

  * Serum creatinine above normal limits ( defined as >500mmol/L)

    * Need for renal replacement therapy
    * History of allergy to study antibiotic
    * Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU with septic shock treated with the study drugs, initiated at the discretion of the treating doctor.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC 0-8h) | Seven blood samples of 3 ml at T0 (pre dose), 30, 45, 60, 120, 240 and 480 mins post infusion completion.
  The concentration versus time data for meropenem & ciprofloxacin in plasma will be analysed by a non-linear mixed effects modelling approach using NONMEM (Version 7.3, GloboMax LLC, Hanover, MD, USA) with double precision with the COMPAQ VISUAL FORTRAN compiler

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Sjoevall, MD, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Sjovall F, Alobaid AS, Wallis SC, Perner A, Lipman J, Roberts JA. Maximally effective dosing regimens of meropenem in patients with septic shock. J Antimicrob Chemother. 2018 Jan 1;73(1):191-198. doi: 10.1093/jac/dkx330. PMID 28961812